CLINICAL TRIAL: NCT03906526
Title: A Phase 1b Multicenter Pre-Surgical Study to Evaluate Immune Biomarker Modulation in Response to Motolimod (VTX-2337) in Combination With Nivolumab in Subjects With Resectable Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: A Study to Evaluate Immune Biomarker Modulation in Response to VTX-2337 in Combination With an Anti- PD-1 Inhibitor in Head and Neck Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VTX-2337-HN-001; U1111-1223-3488 (Registry Identifier: WHO)
Record Dates: First submitted 2018-12-05; First posted 2019-04-08 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Carcinoma, Squamous Cell
Keywords: Motolimod; Nivolumab; Head and Neck Cancer; Squamous Cell Carcinoma; Checkpoint inhibitor; anti-PD1 inhibitor; TLR 8 agonist
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms | interventions — VTX-2337; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Monotherapy Arm 1: Nivolumab (Experimental): Nivolumab IV every 2 weeks
  Interventions: Drug: Nivolumab
- Monotherapy Arm 2: Motolimod (Experimental): Motolimod IT injection weekly
  Interventions: Drug: VTX-2337
- Combination Arm 3: Nivolumab and Motolimod (Experimental): Nivolumab IV every 2 weeks and Motolimod IT injection weekly
  Interventions: Drug: VTX-2337; Drug: Nivolumab
- Combination Arm 4: Nivolumab and Motolimod (Experimental): Nivolumab IV every 2 weeks and Motolimod SC injection weekly
  Interventions: Drug: VTX-2337; Drug: Nivolumab

INTERVENTIONS:
Drug: VTX-2337 — Motolimod
  Other Names: VTX-378
  Arms: Combination Arm 3: Nivolumab and Motolimod; Combination Arm 4: Nivolumab and Motolimod; Monotherapy Arm 2: Motolimod
Drug: Nivolumab — IV Nivolumab
  Other Names: Opdivo
  Arms: Combination Arm 3: Nivolumab and Motolimod; Combination Arm 4: Nivolumab and Motolimod; Monotherapy Arm 1: Nivolumab

SUMMARY:
This is an open label, Phase 1b pre-operative window of opportunity biomarker trial to analyze the combination of intravenous (IV) anti-PD-1 inhibitor, nivolumab, given along with toll-like receptor 8 (TLR 8) agonist motolimod delivered either subcutaneously (SC) or by intratumoral injection (IT) in subjects with squamous cell carcinoma of the head and neck (SCCHN). Subjects with previously untreated, resectable SCCHN, will be recruited onto this trial and will initially undergo pre-treatment diagnostic imaging and biological sample collection. These subjects will undergo pre-operative study treatment for a 3 to 4-week period prior to a scheduled surgical resection.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age at the time of signing the informed consent form (ICF).
* Subject has Eastern Cooperative Oncology Group (ECOG) PS of 0 or 1.
* Subject has a new clinical or pathologic diagnosis of resectable HPV+ or HPV- SCCHN of the oral cavity, pharynx, or larynx
* Macroscopic complete resection of the primary tumor must be planned and subjects should have no medical contraindication to surgery.
* Subject consents to and has tumor accessible for tumor biopsy pre-treatment.
* Subjects must have acceptable hematopoietic, liver, renal, and coagulation function as assessed by laboratory tests.

Exclusion Criteria:

* Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
* Subject has unresectable or inoperable tumors
* Subject has primary tumors of the sinuses, paranasal sinuses, or nasopharynx, or unknown primary tumors
* Subject has evidence of distant metastasis
* Subject is a pregnant or nursing female.
* Subject has active or uncontrolled infection including known HIV infection or known chronic hepatitis B or C.
* Subject has active autoimmune disease.
* Subject has clinically significant ophthalmologic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2022-01-24 (Actual); Study Completion 2022-01-24 (Actual)

PRIMARY OUTCOMES:
Numbers of CD8+ T cells within the tumor pre-treatment and post-surgery | Screening through Study Day 52
  Tumor immune modulation will be evaluated by counting the number of tumor infiltration CD8+ T cells before and after treatment.

SECONDARY OUTCOMES:
Number of Patients With adverse events that lead to delay in resection | Screening through Study Day 52
  Study will evaluate the number of patients who experience adverse events that lead to a significant delay in surgical resection.
Evaluation of safety and tolerability of nivolumab, motolimod and the combination of nivolumab with motolimod | Up to approximately 112 days
  Subject will be monitored for AEs both during treatment and for a specified period after last dose of study treatment. AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (i.e., any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (12):
- United States (12):
  - Local Institution - 112, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Boston University, Boston, Massachusetts
  - Local Institution - 116, Boston, Massachusetts
  - Local Institution - 102, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Local Institution - 101, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Local Institution - 103, Sioux Falls, South Dakota
  - Sanford Cancer Center, Sioux Falls, South Dakota

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome